CLINICAL TRIAL: NCT01889472
Title: Impact of Nasal Mask/Oronasal Mask on Compliance to Treatment With Continuous Positive Airway Pressure (CPAP) in Patients With Obstructive Sleep Apnea
Brief Title: Impact of Interface With/Without Oral Appliance of Sleep Apnea Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to further include additional patients
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Frédéric Sériès, Director IUCPQ sleep laboratory, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MNB-003; JDBF-2012 (Other Grant/Funding Number: JD Begin foundation)
Record Dates: First submitted 2013-06-19; First posted 2013-06-28 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP compliance; leaks; Respiratory disturbances index; quality of life
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oro-nasal mask (Active Comparator): Oro-nasal mask during 1 month of auto CPAP
  Interventions: Device: Nasal mask and oral appliance vs oro-nasal mask during autoCPAP therapy
- Nasal mask and oral appliance (Experimental): Nasal mask and oral appliance during 1 month of auto CPAP
  Interventions: Device: Nasal mask and oral appliance vs oro-nasal mask during autoCPAP therapy

INTERVENTIONS:
Device: Nasal mask and oral appliance vs oro-nasal mask during autoCPAP therapy

SUMMARY:
CPAP is the most effective treatment of obstructive sleep apnea. Oro-nasal masks may be used in case of mouth leaks but these are associated with higher positive pressure needs and lower compliance to treatment. The present investigation evaluates if CPAP compliance would increase when an oral appliance is used in combination with a nasal mask compared to the use of an oro-nasal mask. Eligible patients are those demonstrating a low compliance when using an oro-nasal mask during CPAP therapy. Patients will be treated with automatic CPAP with one of the above-detailed interfaces for 4 weeks and data will be extracted from the machine report in each condition.

DETAILED DESCRIPTION:
Participating subjects will be currently treated by CPAP and low compliance will be assessed according to machine report download demonstrating 3h or less of CPAP usage per night.

ELIGIBILITY:
Inclusion Criteria:

* normal nasal breathing
* dentition allowing for use of an oral appliance
* absence of mandibular joint pathology
* Patients requiring the use of a facial mask during CAPP titration due to presence of mouth leaks with a nasal/prong interface
* Patients using CPAP less than 3 hours/day as prescribed following CPAP titration

Exclusion Criteria:

* Clinical instability
* smoking cessation
* current weight loss strategy
* Marked anatomic abnormalities of upper airway (i.e. macroglossia, tonsils hypertrophy)
* severe cardio-metabolic co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
CPAP compliance | After 4 weeks of CPAP trial
  CPAP compliance will be assessed according to machine report download for the 4 weeks of treatment in each study condition.

SECONDARY OUTCOMES:
diurnal somnolence | After 4 weeks of CPAP trial
  Epworth Sleepiness Score

OTHER OUTCOMES:
Respiratory disturbances index | After 4 weeks of CPAP trial
  Provided by CPAP report

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Series, MD, Principal Investigator — Fondation IUCPQ
Locations (3):
- Canada (2):
  - CHUM, Montreal, Quebec
  - IUCPQ, Québec
- AGIRADOM, Grenoble, France

REFERENCES:
- [Background] Borel JC, Tamisier R, Dias-Domingos S, Sapene M, Martin F, Stach B, Grillet Y, Muir JF, Levy P, Series F, Pepin JL; Scientific Council of The Sleep Registry of the French Federation of Pneumology (OSFP). Type of mask may impact on continuous positive airway pressure adherence in apneic patients. PLoS One. 2013 May 15;8(5):e64382. doi: 10.1371/journal.pone.0064382. Print 2013. PMID 23691209
- [Derived] Leotard A, Lesgoirres M, Daabek N, Lebret M, Bailly S, Verain A, Series F, Pepin JL, Borel JC. Adherence to CPAP with a nasal mask combined with mandibular advancement device versus an oronasal mask: a randomized crossover trial. Sleep Breath. 2019 Sep;23(3):885-888. doi: 10.1007/s11325-018-01772-5. Epub 2019 Jan 28. PMID 30689098